CLINICAL TRIAL: NCT05156203
Title: A Phase I Study of Safety, Tolerability and Pharmacokinetics of T-1301 Capsules in Subjects with Advanced Solid Tumors
Brief Title: Safety and Tolerability Study for T-1301 Capsules to Treat Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taivex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAI-301
Record Dates: First submitted 2021-11-26; First posted 2021-12-14 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- T-1301 Capsules (Experimental): T-1301 Capsules will be administered orally QD or BID in a 28-day cycle (21 days on treatment followed by 7 days off treatment) in sequential cohorts.
  Interventions: Drug: T-1301 Capsules

INTERVENTIONS:
Drug: T-1301 Capsules — T-1301 Capsules, 10 and 50 mg, are opaque hard gelatin capsules for oral administration.

SUMMARY:
T-1301 is a novel small-molecule inhibitor of multiple kinases being developed as an oral drug for the treatment of advanced solid tumors. The nonclinical study results demonstrate the nonclinical efficacy and safety of T-1301 and support the design of this Phase 1, first-in-human (FIH) clinical trial in subjects with advanced cancer.

This study is an open-label, multi-center, Phase I dose-escalation study to evaluate the safety, tolerability, and pharmacokinetics of T-1301 capsules in subjects with advanced solid tumors (including lymphoma), and to identify the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D). Approximately 30 patients will be enrolled for the dose-escalation phase. Actual number of patients will be determined by the number of dose cohorts until the MTD is reached.

T-1301 will be administered orally QD or BID in a 28-day cycle (21 days on treatment followed by 7 days off treatment) in sequential cohorts. Subjects can continue with the treatment until one of the discontinuation criteria is met or until the planned stop of the study (12 months after the last subject receives the first dose of study drug), whichever comes first.

The planned dose levels are: 10, 20, 40, 60, 80, 100, 120, 140 and 160 mg/day. The dosing schedule will be once daily (QD) at the first dose level (10 mg/day) and be changed to twice daily (BID) starting with the second dose level. Other dose levels or dosing frequency may be explored based on safety and related drug exposure data following the decision of Safety Review Committee.

The dose escalation will follow accelerated titration and the Bayesian optimal interval (BOIN) design. During the initial accelerated titration phase, one (1) subject is enrolled per dose level. In the subsequent phase when the BOIN design is used, subjects will be enrolled in cohorts of size 3-6.

ELIGIBILITY:
Inclusion Criteria:

1. Having signed and dated informed consent form indicating that the subject has been informed of all pertinent aspects of the study.
2. Subjects with histologically and cytologically confirmed advanced solid tumors (including lymphoma) that are refractory to standard treatments, or for whom no standard treatment is available, or who are not amenable or unwilling to receive standard treatments.
3. Solid tumors that are measurable or evaluable per Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Target lesions that have been previously irradiated will not be considered measurable (lesion) unless increase in size is observed following completion of radiation therapy.
4. Have a life expectancy of ≥ 3 months in the Investigator's opinion.
5. Females or males ≥ 20 years old.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Recovered from prior treatment-related toxicity to at least grade 1 with the exception of alopecia.
8. Adequate organ function as defined by the following criteria:

   1. Serum alanine transaminase (ALT) ≤ 3 x upper limit of normal (ULN)
   2. Total serum bilirubin ≤ 1.5 x ULN
   3. Absolute neutrophil count (ANC) ≥ 1500/µL
   4. Platelets ≥ 100,000/µL
   5. Hemoglobin ≥ 9.0 g/dL
   6. Creatinine clearance (CrCl) ≥ 50 mL/min CrCl = [(140 - age (year)) x weight (kg)] / (serum creatinine x 72) (x 0.85 for females)
9. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

1. Major surgery within 4 weeks prior to the first dose of study drug.
2. Subjects receiving any of the following anti-cancer therapy:

   1. Anti-cancer definitive radiation therapy (4,000-6,000 cGy) within 4 weeks prior to the first dose of study drug.
   2. Palliative radiation (≤ 10 fractions with total dose < 3,000 cGy) within 2 weeks prior to the first dose of study drug.
   3. Any systemic cytotoxic chemotherapy within 4 weeks prior to the first dose of study drug.
   4. Any targeted therapy within 2 weeks or 5 half-lives, whichever is longer, prior to the first dose of study drug.
   5. Any immunotherapy within 4 weeks prior to the first dose of study drug.
3. Any interventional treatments in another clinical trial following Exclusion Criteria 2c, 2d and 2e.
4. Subjects received blood transfusion or biological response modifiers (e.g., G-CSF) within 2 weeks prior to the first dose of study drug.
5. Subject who received autologous bone marrow transplant or stem cells rescue within 6 months prior to the first dose of study drug.
6. Subjects received strong inhibitors and/or inducers of CYP3A4 within 14 days prior to the first dose of study drug. A list of CYP3A4 modulators is provided in Appendix 3.
7. Documented or suspected brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease.
8. Any of the following within 6 months of the first dose of study drug: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack.
9. Ongoing cardiac dysrhythmias of ≥ NCI CTCAE version 5.0 grade 2, or atrial fibrillation of any grade. Corrected QT interval by Fridericia (QTcF) ≥ 470 msec.
10. Hypertension that cannot be controlled by medications (> 160/100 mm-Hg despite optimal medical therapy).
11. AIDS-defining opportunistic infections within the past 12 months.
12. Positive test for hepatitis B (HBsAg) or hepatitis C (anti-HCV (anti-hepatitis C virus) antibody), unless the HCV RNA level is below the limit of detection (for subjects with positive anti-HCV Ab).
13. Men and women of childbearing potential who are unwilling to use highly effective contraceptive methods during the study period.

    Highly effective contraceptive methods include implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, surgical sterilization or a partner who is sterile.
14. If females, patient is pregnant or breast feeding.
15. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart, in the judgement of the investigator and/or sponsor, excess risk associated with study participation or study drug administration.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | First treatment cycle (i.e., the first 28 days post the first dose)
  The MTD will be selected based on isotonic regression as specified in Liu and Yuan (2015). Specifically, the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate is selected as the MTD. If there are ties, the higher dose level is selected when the isotonic estimate is lower than the target toxicity rate and the lower dose level is selected when the isotonic estimate is greater than or equal to the target toxicity rate. The target toxicity rate for the MTD is 30% and the MTD will be determined based on the occurrence of the dose-limiting toxicity (DLT) assessed using toxicity data during Cycle 1 (the first 28 days).
Recommended phase 2 dose (RP2D) | First treatment cycle (i.e., the first 28 days post the first dose)
  The recommended Phase 2 Dose (RP2D) will not exceed the MTD and will be determined by the Safety Review Committee.
Frequency, types, severity and relationship to study drug of adverse events (AEs) | At least 84 days (i.e., 56 days for two treatment cycles and 28 days for safety follow-up)
  Safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Cmax | Selected time points during the first 28-day treatment cycle
  The maximum plasma concentration of T-1301 derived from the plasma concentration-time profiles
Pharmacokinetic parameters: Ctrough | Selected time points during the first 28-day treatment cycle
  The plasma concentration of T-1301 at trough level derived from the plasma concentration-time profiles
Pharmacokinetic parameters: Tmax | Selected time points during the first 28-day treatment cycle
  The time to reach maximum concentration of T-1301 derived from the plasma concentration-time profiles
Pharmacokinetic parameters: AUC | Selected time points during the first 28-day treatment cycle
  The area under the concentration versus time curve of T-1301 derived from the plasma concentration-time profiles
Pharmacokinetic parameters:T1/2 | Selected time points during the first 28-day treatment cycle
  The terminal half-life of T-1301 derived from the plasma concentration-time profiles.
Objective response rate (ORR) | At least 56 days
  To assess preliminary anti-tumor activity with ORR according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - ChangGung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided